CLINICAL TRIAL: NCT02852733
Title: Better Understand End-of-life Emergencies' Management Among Elderly in Nursing Homes: a Pilot Study in Brittany, France
Acronym: PUFPAE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC12_8988
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Died; in End-of-life Situation
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (2):
- Residents in end-of-life situation: Residents in end-of-life situation the day of the survey, as determined by the physician coordinator of nursing homes (we will use the definition of "terminal condition" contained in the guide of the CNSA (coding PATHOS - April 2011)).
  Interventions: Other: end-of-life emergencies' management
- dead residents: dead residents in the quarter preceding the date of the survey
  Interventions: Other: end-of-life emergencies' management

INTERVENTIONS:
Other: end-of-life emergencies' management

SUMMARY:
The purposes of this study are :

* To know and to understand frequency and variability (quantitative and qualitative) of end-of-life emergencies in nursing homes.
* To know and to understand practices applied in these situations depending on the institution and the different reasons of hospital use.
* To know and to understand the practical and organizational elements, in nursing homes, that can determine a (re) hospitalization or an end-of-life

ELIGIBILITY:
Inclusion Criteria:

* dead residents during the quarter preceding the date of the Survey Or
* Residents in end-of-life situation the day of the survey, as determined by the physician coordinator of nursing homes (we will use the definition of "terminal condition" contained in the guide of the CNSA (coding PATHOS - April 2011)).

Exclusion Criteria:

* patients opposing the study,
* patients aged below 18 year old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Résidents of 150 nursing homes randomly selected in Brittany
Sampling Method: Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
number of end-of-life emergencies' episodes | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francoise FR RIOU, MD, Study Director — Rennes University Hospital
Locations (1):
- CHU de RENNES, Rennes, France